CLINICAL TRIAL: NCT05785585
Title: Effect of Methylcobalamin and Cyanocobalamin Consumption on Vitamin B12 Nutritional Status in Vegetarians With Marginal Vitamin B12 Deficiency. Randomized, Parallel, Placebo-Controlled, Triple-Blind Clinical Trial.
Brief Title: Effect of Methylcobalamin and Cyanocobalamin Consumption on Vitamin B12 Nutritional Status
Acronym: NORMB12
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Eurecat (Other)
Collaborators: Laboratorio Echevarne (Industry); Health Tech Bio Actives, S.L.U. (Unknown)
Responsible Party: Principal Investigator, Antoni Caimari, Director of Eurecat's Biotechnology Area, Principal Investigator, Fundació Eurecat
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NORMB12
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Vitamin B12 Nutritional Deficiency
Keywords: Vitamin B12; Methylcobalamin; Cyanocobalamin; Vegetarians; Holotranscobalamin; Methylmalonic acid; Homocysteine; 4cB12
MeSH Terms: interventions — mecobalamin; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Methylcobalamin group (Experimental): One capsule daily with 500 µg of methylcobalamin for 12 weeks
  Interventions: Dietary Supplement: Methylcobalamin
- Cyanocobalamin group (Active Comparator): One capsule daily with 500 µg of Cyanocobalamin for 12 weeks
  Interventions: Dietary Supplement: Cyanocobalamin group
- Control group (Placebo Comparator): One capsule daily with microcrystalline cellulose for 12 weeks
  Interventions: Dietary Supplement: Control group

INTERVENTIONS:
Dietary Supplement: Methylcobalamin — Treatment with Methylcobalamin during 12 weeks
  Arms: Methylcobalamin group
Dietary Supplement: Cyanocobalamin group — Treatment with Cyanocobalamin during 12 weeks
  Arms: Cyanocobalamin group
Dietary Supplement: Control group — Treatment with microcrystalline cellulose during 12 weeks
  Arms: Control group

SUMMARY:
Vitamin B12 (B12, Cobalamin) is an essential micronutrient that humans are not capable of synthesizing and therefore must be ingested through food. In nature, B12 is basically only present in foods of animal origin.

B12 deficiency is a clinically important condition that is associated with several metabolic disorders such as megaloblastic anemia, hyperhomocysteinemia, and cardiovascular, cerebrovascular, and neurological disorders. Therefore an optimal intake of B12 is important.

B12 deficiency occurs when B12 stores are depleted due to inadequate dietary intake or impaired absorption of B12. Because B12 is only present in foods of animal origin, following an unbalanced vegetarian diet is associated with increased risk of developing nutritional deficiencies due to the exclusion of meat and fish from their diet, including vitamin B12 deficiency.

There are a variety of forms of vitamin B12 used in vitamin B12 supplements. All these forms share the structure of Cobalamin but contain different ligands. Cyanocobalamin (CNCbl) is a synthetic, stable, and inexpensive form widely used in B12 supplements. MethylCobalamin (MeCbl) is a physiological form of cobalamin, called metabolically active form of vitamin B12. Interest in substituting CNCbl form with the physiological form MCbl has recently increased, assuming that it will be more effective.

The main objective of the study is to evaluate the effect of Methylcobalamin consumption, compared to Cyanocobalamin consumption, on the nutritional status of vitamin B12 in a vegetarian population with marginal vitamin B12 deficiency.

The secondary objectives of the study are to evaluate the effects of Methylcobalamin consumption, compared to Cyanocobalamin consumption, on markers of vitamin B12 deficiency: Holotranscobalamin, Methylmalonic acid, Homocysteine and 4cB12.

During the study there will be 8 visits: a preselection visit (V0; day -7) and 7 study visits during the consumption of the treatments, which will take place on the first day of the study (V1; day 1), after 8 days of treatment (V2; day 8), at 15 days of treatment (V3; day 15), at 29 days of treatment (V4; day 29), at 43 days of treatment (V5; day 43), at 64 days of treatment (V6; day 64), and at 85 days of treatment (V7; day 85).

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years or older who follow a vegetarian diet.
* Present serum vitamin B12 levels of 148-221 pmol/L and absence of symptoms associated with vitamin B12 deficiency.
* Sign the informed consent.
* Read, write and speak Catalan or Spanish.

Exclusion Criteria:

* Present diagnosed diseases that may interfere with vitamin B12 markers, including gastrointestinal diseases (such as inflammatory bowel disease, celiac disease, ileal resection, Crohn's disease, constipation or atrophic gastritis), pancreatic diseases, kidney diseases, liver diseases, diabetes, cardiovascular diseases, pernicious anemia and cancer.
* Medical history of abdominal surgery that may influence the absorption of vitamin B12 (such as bariatric surgery).
* Being on hemodialysis treatment.
* Present values of body mass index ≤ 18.5 kg/m^2 or ≥ 35 kg/m^2.
* Present anemia (hemoglobin ≤ 13 g/dL in men and ≤ 12 g/dL in women).
* Having consumed or consume vitamin B12 or folate supplements for more than 2 months before inclusion in the study.
* Have taken medications that affect the absorption and therapeutic response of vitamin B12 (such as methotrexate, metformin, proton pump inhibitors, H2 receptor antagonists, histamine, nitrous oxide, colchicine, neomycin, biguanides, cholestyramine, aminosalicylic acid, chloramphenicol and other bone marrow depressants) one month before inclusion in the study.
* Be a smoker or ex-smoker in the last 6 months before inclusion in the study.
* Take 2 or more Standard Beverage Units (SBU) daily or 17 SBU weekly for women, or take 4 or more SBU daily or 28 SBU weekly for men.
* Present allergy or intolerance to the study products (microcrystalline cellulose, vitamin B12 or cobalt).
* Being pregnant or intending to become pregnant.
* Being in breastfeeding period.
* Participate in or have participated in a clinical trial or nutritional intervention study in the last 30 days before inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-09-09 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Levels of total vitamin B12 in blood. | At day -7 (pre-selection visit), day 8 (visit 2), day 15 (visit 3), day 29 (visit 4), day 43 (visit 5), day 64 (visit 6) and day 85 (visit 7).
  Serum total vitamin B12 will be measured by chemiluminescence immunoassay.

SECONDARY OUTCOMES:
Levels of Holotranscobalamin in blood. | At day -7 (pre-selection visit), day 8 (visit 2), day 15 (visit 3), day 29 (visit 4), day 43 (visit 5), day 64 (visit 6) and day 85 (visit 7).
  Serum Holotranscobalamin will be measured by chemiluminescence immunoassay.
Levels of Methylmalonic acid in blood. | At day -7 (pre-selection visit), day 8 (visit 2), day 15 (visit 3), day 29 (visit 4), day 43 (visit 5), day 64 (visit 6) and day 85 (visit 7).
  Serum Methylmalonic acid will be measured by Liquid Chromatography coupled to tandem Mass Spectrometry.
Levels of Homocysteine in blood. | At day -7 (pre-selection visit), day 8 (visit 2), day 15 (visit 3), day 29 (visit 4), day 43 (visit 5), day 64 (visit 6) and day 85 (visit 7).
  Plasma Homocysteine will be measured by Liquid Chromatography coupled to tandem Mass Spectrometry.
Levels of 4cB12 marker. | At day -7 (pre-selection visit), day 8 (visit 2), day 15 (visit 3), day 29 (visit 4), day 43 (visit 5), day 64 (visit 6) and day 85 (visit 7).
  The 4cB12 marker will be calculated from the blood levels obtained for total vitamin B12, Holotranscobalamin, Methylmalonic acid and Homocysteine using the formula log10((B12 x Holotranscobalamin)/(Methylmalonic acid x Homocysteine)).
Levels of folate in blood. | At day -7 (pre-selection visit) and day 85 (visit 7).
  Serum folate will be measured by chemiluminescence immunoassay.
Levels of vitamin B6 in blood. | At day -7 (pre-selection visit) and day 85 (visit 7).
  Plasma vitamin B6 will be measured by Ultra High Performance Liquid Chromatography coupled to tandem Mass Spectrometry.
Health related quality of life. | At day 1 (visit 1) and day 85 (visit 7).
  Health related quality of life will be assessed using the SF-36 questionnaire (36-item short form survey) in Spanish. The SF-36 questionnaire consists of the subscales general health (5 items), mental health (5 items), emotional role (3 items), social function (2 items), vitality (4 items), physical function (10 items), physical role (4 items) and bodily pain (2 items). The items on the scale are ordered in such a way that the higher the score, the higher the state of health. Scores on each of the SF-36 scales range from 0 to 100.
Dietary habits and caloric intake. | At day 1 (visit 1) and day 85 (visit 7).
  Nutritional habits and caloric intake will be determined based on the results obtained from the 3-day dietary record.
Consumption of foods with vitamin B12. | At day 1 (visit 1), day 8 (visit 2), day 15 (visit 3), day 29 (visit 4), day 43 (visit 5), day 64 (visit 6) and day 85 (visit 7).
  Consumption of foods with vitamin B12 by the volunteers will be determined by analyzing the questionnaire on the frequency of consumption of foods with vitamin B12.
Compliance with dietary recommendations. | At day 8 (visit 2), day 15 (visit 3), day 29 (visit 4), day 43 (visit 5), and day 64 (visit 6).
  The adherence to the dietary recommendations by the volunteers will be determined by analyzing the 24h dietary recall.
Physical activity. | At day 1 (visit 1) and day 85 (visit 7).
  Physical activity will be evaluated through the International Physical Activity Questionnaire (IPAQ)-short for physical activity questionnaire.
Concomitant medication. | At day 1 (visit 1), day 8 (visit 2), day 15 (visit 3), day 29 (visit 4), day 43 (visit 5), day 64 (visit 6) and day 85 (visit 7).
  The consumption of concomitant medication by te volunteers will be controlled by the record of concomitant medication in the case report form.
Consumption of food supplements. | At day 1 (visit 1), day 8 (visit 2), day 15 (visit 3), day 29 (visit 4), day 43 (visit 5), day 64 (visit 6) and day 85 (visit 7).
  The consumption of food supplements by te volunteers will be controlled by the record of food supplements in the case report form.
Body weight. | At day 1 (visit 1) and day 85 (visit 7).
  Body weight measured by standardized method.
Height. | At day -7 (pre-selection visit).
  Height measured by standardized method.
Body Mass Index. | At day 1 (visit 1) and day 85 (visit 7).
  Weight and height will be combined to report Body Mass Index in kg/m^2.
Age. | At day -7 (pre-selection visit).
  The age of the volunteers will be recorded in the case report form.
Gender. | At day -7 (pre-selection visit).
  The gender of the volunteers will be recorded in the case report form.
Intervention compliance. | At day 43 (visit 5) and day 85 (visit 7).
  The intervention compliance by te volunteers will be assessed by counting the number of remaining capsules and applying the formula (Number of capsules consumed/Number of capsules to consume)x100.
Adverse events. | At day 8 (visit 2), day 15 (visit 3), day 29 (visit 4), day 43 (visit 5), day 64 (visit 6) and day 85 (visit 7).
  Possible adverse events derived from taking study's products will be recorded in the case report form.

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Caimari, PhD, Principal Investigator — Fundació Eurecat
Locations (2):
- Spain (2):
  - Fundació Eurecat, Reus, Tarragona
  - Eurecat, Reus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Technological Centre of Nutrition and Health. Eurecat_Reus. — http://eurecat.org